CLINICAL TRIAL: NCT01917916
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Doses of BI 655064 (Buffer Solution for Injection) in Healthy Chinese and Japanese Male Volunteers (Randomised, Double-blind, Placebocontrolled Within Dose Groups, Clinical Phase I Study)
Brief Title: Single Rising Doses of BI 655064 in Healthy Chinese and Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1293.8
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — BI 655064

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- BI 655064 dose group 1 - 80 mg (Experimental)
  Interventions: Drug: BI 655064
- BI 655064 dose group 2 - 120 mg (Experimental)
  Interventions: Drug: BI 655064
- BI 655064 dose group 3 - 180 mg (Experimental)
  Interventions: Drug: BI 655064
- BI 655064 dose group 4 - 240 mg (Experimental)
  Interventions: Drug: BI 655064
- Placebo matching BI 655064 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Solution for subcutaneous (s.c.) injection.
  Arms: Placebo matching BI 655064
Drug: BI 655064 — Solution for subcutaneous (s.c.) injection.
  Arms: BI 655064 dose group 1 - 80 mg; BI 655064 dose group 2 - 120 mg; BI 655064 dose group 3 - 180 mg; BI 655064 dose group 4 - 240 mg

SUMMARY:
Safety, tolerability, pharmacokinetics and pharmacodynamics of BI 655064 after single rising doses in healthy Asian male volunteers.

ELIGIBILITY:
Inclusion criteria:

* Healthy males based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Chinese ethnicity, Japanese ethnicity according to the following criteria. Japanese: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan. Chinese: ethnic Chinese, born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
* Age within the range of 20 to 45 years inclusive
* Body mass index within the range of 18.5 and 25 kg/m2 inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any disease or clinically relevant abnormality in laboratory parameters which, according to the investigator, might compromise the safety of the subject or interfere with the subjects participation in the trial or compromise the trial objectives
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2014-05-14 (Actual); Study Completion 2014-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- 1293.8.8101 Boehringer Ingelheim Investigational Site, Sumida-ku,Tokyo, Japan
- 1293.8.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind within dose groups, single rising dose study with 4 doses in Chinese and Japanese healthy volunteers.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 655064 Dose Group 1 - 80 mg: Japanese and Chinese healthy participants were administered subcutaneously (s.c.) a single dose of 80 milligram (mg) of solution for injection of BI 655064.
- BI 655064 Dose Group 2 - 120 mg: Japanese and Chinese healthy participants were administered subcutaneously (s.c.) a single dose of 120 milligram (mg) of solution for injection of BI 655064.
- BI 655064 Dose Group 3 - 180 mg: Japanese and Chinese healthy participants were administered subcutaneously (s.c.) a single dose of 180 milligram (mg) of solution for injection of BI 655064.
- BI 655064 Dose Group 4 - 240 mg: Japanese and Chinese healthy participants were administered subcutaneously (s.c.) a single dose of 240 milligram (mg) of solution for injection of BI 655064.
- Placebo Matching BI 655064: Japanese and Chinese healthy participants were administered subcutaneously (s.c.) a single dose of solution for injection of Placebo matching BI 655064.
Period: Overall Study
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg | Placebo Matching BI 655064
Started | 12 | 12 | 12 | 12 | 16
Completed | 12 | 12 | 12 | 12 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set included all subjects who were documented to have taken study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg | Placebo Matching BI 655064 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (6.7) | 24.6 (2.6) | 26.7 (6.0) | 29.7 (9.7) | 26.1 (5.6) | 26.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 12 | 12 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator Defined Drug-related Adverse Events
Description: Number of participants with investigator defined drug-related adverse events (AEs) is reported.
Time Frame: From study drug administration until end-of-study examination, up to 77 days.
Population: Treated Set (TS): This subject set included all subjects who were documented to have taken study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg | Placebo Matching BI 655064
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 16
Participants | 2 | 1 | 4 | 2 | 1

2. Secondary Outcome: Maximum Measured Concentration of BI 655064 in Plasma (Cmax)
Description: Maximum measured concentration of BI 655064 in plasma (Cmax) is reported.
Time Frame: Within 3:00 hours:minutes (h:min) before and 08:00h, 12:00h, 24:00h, 36:00h, 48:00h, 72:00h, 96:00h, 108:00h, 120:00h, 168:00h, 264:00h, 432:00h, 648:00h, 984:00h, 1320:00h, 1656:00 h:min after BI 655064 administration.
Population: The pharmacokinetic (PK) set (PKS) included all subjects from the treated set (TS) who provided at least 1 secondary PK endpoint that was judged as PK evaluable and was not affected by protocol violations relevant to the statistical evaluation of PK endpoints. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)/ (milliliter) mL
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
nanogram (ng)/ (milliliter) mL
  Chinese participants: number analyzed (Participants) | 6 | 6 | 6 | 6
  Chinese participants | 888 (501) | 5160 (51.6) | 8650 (41.1) | 15700 (54.2)
  Japanese participants: number analyzed (Participants) | 5 | 6 | 6 | 6
  Japanese participants | 1550 (315) | 7210 (92.8) | 16300 (73.6) | 21300 (53.4)
Statistical Analysis 1: Comparison: BI 655064 Dose Group 1 - 80 mg vs BI 655064 Dose Group 2 - 120 mg vs BI 655064 Dose Group 3 - 180 mg vs BI 655064 Dose Group 4 - 240 mg; Dose proportionality was explored using the power model. Dose proportionality of BI 655064 was to be assessed based on the exposure parameter Cmax, determined for the 4 subcutaneous dose levels. This analysis is for the overall population; Test type: Other; Slope = 2.4386, 95% CI 2-sided [1.7504 to 3.1267], Standard Error of Mean 0.3417 — Perfect dose proportionality would correspond to a slope of 1. Standard error of mean is actually standard error of slope

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI 655064 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte BI 655064 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is reported.
Time Frame: as for outcome 2
Population: The pharmacokinetic (PK) set (PKS) included all subjects from the treated (TS) who provided at least 1 secondary PK endpoint that was judged as PK evaluable and was not affected by protocol violations relevant to the statistical evaluation of PK endpoints. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)*hours (h)/mL
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg
Number analyzed (Participants) | 10 | 12 | 12 | 11
microgram (µg)*hours (h)/mL
  Chinese participants: number analyzed (Participants) | 5 | 6 | 6 | 5
  Chinese participants | 330 (111) | 1120 (46.6) | 2910 (60.1) | 5610 (59.0)
  Japanese participants: number analyzed (Participants) | 5 | 6 | 6 | 6
  Japanese participants | 464 (74.1) | 2020 (78.8) | 6430 (83.3) | 7780 (57.1)
Statistical Analysis 1: Comparison: BI 655064 Dose Group 1 - 80 mg vs BI 655064 Dose Group 2 - 120 mg vs BI 655064 Dose Group 3 - 180 mg vs BI 655064 Dose Group 4 - 240 mg; Dose proportionality was explored using the power model. Dose proportionality of BI 655064 was to be assessed based on the exposure parameter AUC0-∞, determined for the 4 subcutaneous dose levels. This analysis is for the overall population; Test type: Other; Slope = 2.6033, 95% CI 2-sided [2.0993 to 3.1073], Standard Error of Mean 0.2499 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte BI 655064 in the Plasma Over the Time Interval From 0 to the Last Measurable Time Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte BI 655064 in the plasma over the time interval from 0 to the last measurable time point (AUC0-tz) is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)*hours (h)/mL
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg
Number analyzed (Participants) | 11 | 12 | 12 | 12
microgram (µg)*hours (h)/mL
  Chinese participants: number analyzed (Participants) | 6 | 6 | 6 | 6
  Chinese participants | 126 (1740) | 1110 (47.2) | 2900 (60.4) | 5680 (52.4)
  Japanese participants: number analyzed (Participants) | 5 | 6 | 6 | 6
  Japanese participants | 365 (165) | 2010 (79.8) | 6380 (84.6) | 7750 (57.2)
Statistical Analysis 1: Comparison: BI 655064 Dose Group 1 - 80 mg vs BI 655064 Dose Group 2 - 120 mg vs BI 655064 Dose Group 3 - 180 mg vs BI 655064 Dose Group 4 - 240 mg; Dose proportionality was explored using the power model. Dose proportionality of BI 655064 was to be assessed based on the exposure parameter AUC0-tz, determined for the 4 subcutaneous dose levels. This analysis is for the overall population; Test type: Other; Slope = 3.1291, 95% CI 2-sided [2.3395 to 3.9187], Standard Error of Mean 0.3920 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From study drug administration until end-of-study examination, up to 77 days.
Description: Treated Set (TS): This subject set included all subjects who were documented to have taken study medication.
Arm/Group | BI 655064 Dose Group 1 - 80 mg | BI 655064 Dose Group 2 - 120 mg | BI 655064 Dose Group 3 - 180 mg | BI 655064 Dose Group 4 - 240 mg | Placebo Matching BI 655064
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12 | 5/12 | 4/12 | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655064 Dose Group 1 - 80 mg (N=12) | BI 655064 Dose Group 2 - 120 mg (N=12) | BI 655064 Dose Group 3 - 180 mg (N=12) | BI 655064 Dose Group 4 - 240 mg (N=12) | Placebo Matching BI 655064 (N=16)
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Administration site rash (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.